CLINICAL TRIAL: NCT06095024
Title: INDIGO Community Participant Led Electronic Completion of PROMs and PREMs for Patients Living With and Beyond Cancer in the Community
Brief Title: INvestigating DIGital Outcomes in the Community
Acronym: INDIGO-Com
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 000000
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Linked to national data: Patients will be randomly assigned to be asked to link personal data with national cancer data.
  The outcome measure will be the proportion of completed questionnaires
- Linking to national data, early vs. late questions: Subset of cohort 1: Patients will be randomly assigned to be asked the question about data linkage at the beginning vs. end of the questionnaire
  The outcome measure will be the proportion answering yes in each arm
- Different PROM Completion rate: Patients will be randomised to two different PROM questionnaires
  The outcome measure will be the completion rate of the two different questionnaires
- Impact of additional PROMS on completion and satisfaction: Patients will be randomised to either a standard PROM or additional, symptom directed questionnaire
  The outcome measure will be the satisfaction rate of patients in each arm

SUMMARY:
To explore the feasibility and best methodology for collecting patient-reported outcome measures in patients who have previously been treated for cancer and are living in the community.

The investigators are working with primary care research teams, and using an online electronic questionnaire. Although the study is entirely observational, the study offers some of the questions in a random order, so the investigators can explore the effect of changing the way in which questions are asked.

DETAILED DESCRIPTION:
INDIGO Community aims to both collect data on patient-reported outcome measures (PROMS) and patient-reported experience measures (PREMS) and data on the impact of how to do this.

The focus is on adult patients living in the community who have previously been treated for cancer.

The study uses a range of quality of life questionnaires, and randomises the order in which some questions are asked, in order to explore the impact of how questions are asked on responses.

All patients with be offered the EuroQol 5 dimension, 5 level questionnaire (EQ5D-5L)

ELIGIBILITY:
Inclusion Criteria:

* Anyone over the age of 16 who has been diagnosed (receiving treatment is not an inclusion criteria although the investigators expect as this is a long-term survivorship study all participants will have received treatment) for any type of cancer in the past (> 12 months) can participate.
* Participants who self-identify as having previously (time unlimited) received a diagnosis of cancer, based on histological, radiological, or clinical grounds (primary and/or metastatic cancer). Current treatment is not a barrier to participation, but the emphasis is on patients who have completed treatment.

Participants need to be able to access the secure online platform, using a mobile device or computer.

* Have capacity and be able to provide informed consent via the online platform.
* To be able to understand, read and write English, with or without support from a trusted individual e.g., friends, family, carer.

Exclusion Criteria:

* Participants recently diagnosed with cancer (less than 12 months ago).
* Participants unable to access secure online platform.
* Participants who do not have sufficiently good understanding of written English to complete the PROMs and are unable to be supported by a trusted individual to complete the questionnaire.
* Participants lacking capacity and unable to give informed consent.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All adults living with a previous diagnosis of cancer in a defined geographical area (NW London in stage 1; nationally in stage 2)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Completion of study questionnaire | 12 months
  Proportion of patients completing the entire study questionnaire
Agreement to link to national cancer data | 12 months
  Proportion of patients agreeing to link their data to national cancer data

SECONDARY OUTCOMES:
Completion of PROMs questionnaires | 12 months
  Proportion of patients completing PROMS questionnaires
Satisfaction with questionnaires | 12 months
  Patient-reported satisfaction with questionnaires, expressed as average scores (on a scale of 1 - 10, where 10 is better) and proportion scoring 5 or over
Effectiveness of different communication channels for recruitment | 12 months
  Enrolment rate via different recruitment channels (Primary Care Research Network, Social Media) expressed as the proportion of patient recruited via each channel
Correlation of each PROM score with quality of life | 12 months
  Correlation of each PROM score with the EuroQol 5 Dimensions, 5 levels (EQ5D-5L) quality of life measure

OTHER OUTCOMES:
The feasibility of developing a national longitudinal cohort | 12 months
  To assess what proportion of participants agree to ongoing, long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Williams, MBChB PhD FRCR, Principal Investigator — Imperial College Healthcare Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be shared, where patients give permission, with the national cancer registration service. Future researchers may then access the data via that route.

REFERENCES:
- [Derived] Le Calvez K, Gregory JJ, Gath J, Wheatstone P, Ashley L, Chinembiri O, Cunliffe A, Davenport G, Jamieson Gilmore K, Langel K, Miglio C, Pakzad-Shahabi L, Padmasri D, Ruta D, Williams H, Williams M. INDIGO randomised controlled digital clinical trial: INvestigating DIgital outcomes and quality of life in cancer survivors - a study protocol. BMJ Open. 2025 Sep 8;15(9):e104336. doi: 10.1136/bmjopen-2025-104336. PMID 40921632